CLINICAL TRIAL: NCT03753373
Title: Acupuncture for Medial Tibial Stress Syndrome in the Primary Care Setting: A Randomized Controlled Trial
Brief Title: Acupuncture for Medial Tibial Stress Syndrome in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eglin AFB Regional Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FWH20180168H
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Medial Tibial Stress Syndrome
Keywords: acupuncture; Medial Tibial Stress Syndrome
MeSH Terms: conditions — Medial Tibial Stress Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture and Home Exercise (Experimental): Acupuncture plus the prescribed home exercise program
  Interventions: Other: Acupuncture; Other: Home Exercise Program
- Home Exercise Only (Active Comparator): The prescribed home exercise program alone
  Interventions: Other: Home Exercise Program

INTERVENTIONS:
Other: Acupuncture — Acupuncture treatments will be utilizing the KB-2 points with manual manipulation accomplished by vigorously running the acupuncturists thumb nail up and down the handle until a perceived sensation change is noted in the subject's posteromedial tibia. A single, sterile 100mm needle will be inserted into the upper third of the medial tibiofibular ligament, followed by a second needle approximately 2-4 cm below the second needle. The needles will be manipulated as detailed above to achieve the sensation change along the posteromedial tibia. The needles will then be irregularly stimulated over the course of 5-7 minutes. The needles will be removed after the treatment is complete, which will last approximately 5-10 minutes (standard care).
  Arms: Acupuncture and Home Exercise
Other: Home Exercise Program — Subjects will be given a study diary to document the number of times they performed the standard of care prescribed home exercise program. Subjects will be advised to complete the stretching exercises daily and the strengthening exercises every other day.

SUMMARY:
The investigators want to investigate whether the KB2 acupuncture protocol is an effective method for decreasing pain and improving physical function in adult subjects with medial tibial stress syndrome. The investigators hypothesize that there will be significant improvement in both the acute and long-term timeframes, with respect to measures of pain and function. The investigators will measure shin pain immediately prior to treatment (baseline), immediately after initial treatment, one-, two-, and four-weeks following treatment, then again at three months post-treatment. Functional status will be evaluated at the above intervals using the Pain Disability Index. The Medial Tibial Stress Syndrome (MTSS) Score is a newly developed scoring system for subject-reported outcomes in evaluating treatment of MTSS, and this will be used to evaluate pain relief and physical functional status at initial treatment (baseline) and again at the four-week follow-up. If at the four-week follow-up no significant improvement is noted, subjects in the non-acupuncture treatment group will be given the option to crossover to another KB2 acupuncture treatment regimen, with follow-up as previously noted.

DETAILED DESCRIPTION:
All of the below items are research-related unless marked as 'standard of care':

Screening Visit:

* Obtain and document signed Informed Consent document and HIPAA Authorization.
* Review past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) to verify the inclusion/exclusion criteria including previous encounter, vital signs review, medication list, co-morbidities, demographics, and problems list.
* Record: Date of birth, age, gender, race, ethnicity, DOD ID#, name of standard of care medications (over-the-counter and prescription), current email address (to be used for scheduling), height (in inches), weight (in pounds), tobacco-use status, duration of current shin splints, history of shin splints, and note any prior acupuncture received.
* Investigators will ask what the subjects expectations are regarding acupuncture's effectiveness for medial tibial stress syndrome.
* If the subject is an active duty member, investigators will ask:

  * Have you or are you currently on a fitness restriction for medial tibial stress syndrome.
  * If so, what are the dates of the restriction?
* There are several standard of care treatments and physical therapy options for the treatment of medial tibial stress syndrome which include physical therapy and a home exercise program. Investigators will standardize what patients in this study are receiving by having all subjects follow the standard of care prescribed home exercise program and discontinue any formal physical therapy when entering this study (regular physical activity such as exercise is allowed, as tolerated by pain level).

Randomization: Subjects will be randomized into 1 of 2 equal groups, using a random number generator:

* Group 1: Acupuncture plus the prescribed home exercise program
* Group 2: The prescribed home exercise program alone

Encounter 1--Day 1 (may be same day as screening visit):

* Subjects will be given a study diary to document the number of times they performed the standard of care prescribed home exercise program. Subjects will be advised to complete the stretching exercises daily and the strengthening exercises every other day.
* Self-reported pain severity pre-intervention (0 for no pain to 10 being the worst pain)
* Research treatment intervention according to their randomization group:

  * Group 1:

Acupuncturist will be given a copy of the Protocol for Needle Insertion. Acupuncture will be performed. The name of the physician performing the acupuncture and also the number of acupuncture needles placed for each treatment.

The prescribed home exercise program will be reviewed. o Group 2: The prescribed home exercise program will be reviewed.

* Self-reported pain severity post-intervention (0 for no pain to 10 being the worst pain)
* Administer the Pain Disability Index (PDI), Medial Tibial Stress Syndrome Score (MTSS Score) electronically
* Subjects will be instructed to perform the stretching exercises daily and the strengthening exercises every other day.

Encounter 2-- Week 2 Survey:

• Electronic completion of PDI, MTSS Score, pain scale, and patient reported frequency of home exercise program diary

Encounter 3-- Week 4 Survey:

* Electronic completion of PDI, MTSS Score, pain scale, and patient reported frequency of home exercise program diary.
* Subjects in the non-acupuncture treatment group, with failure of pain scale to decrease by 2 points on 0-10 point pain scale, will be given the option to crossover to the acupuncture treatment group, receive acupuncture, and continue scheduled follow-up at 2, 4, and 12 weeks.

Encounter 4-- Week 12 Survey:

* Electronic completion of PDI, MTSS Score, pain scale, and patient reported frequency of home exercise program diary
* Investigators will ask if the subject's expectations regarding acupuncture's effectiveness for medial tibial stress syndrome were met.

Acupuncture: For purposes of this study, acupuncture will be considered a research-related intervention and all acupuncturists performing the procedure will be considered engaged investigators for research purposes. For this study, all physician acupuncturists are deemed engaged research investigators, since the acupuncture procedure is research-related for the study. Unless the acupuncturist is added to the study, they will not be permitted to perform the acupuncture procedure s on the research subjects. Acupuncture treatments will be utilizing the KB-2 points with manual manipulation accomplished by vigorously running the acupuncturists thumb nail up and down the handle until a perceived sensation change is noted in the subject's posteromedial tibia. A single, sterile 100mm needle will be inserted into the upper third of the medial tibiofibular ligament, followed by a second needle approximately 2-4 cm below the second needle. The needles will be manipulated as detailed above to achieve the sensation change along the posteromedial tibia. The needles will then be irregularly stimulated over the course of 5-7 minutes. The needles will be removed after the treatment is complete, which will last approximately 5-10 minutes (standard care).

Acupuncture treatments will be as defined: KB-2 are generally not defined specific points, but are referred to the placement of the needle into the lateral leg and advanced through the medial tibiofibular ligament (interosseous membrane). The initial KB-2 point will be placed in the upper 1/3 of the leg distal to the tibial tuberosity. The second needle will be placed 2-4 cm below the first needle, still within the upper 1/3 of the leg.

This study will follow all FDA requirements for the safe use of these devices.

The acupuncture being performed in this study is a standard acupuncture technique for the treatment of medial tibial stress syndrome. However, for this study, the research-related acupuncture procedure being performed is considered research-related. The physicians performing the treatment are trained in this acupuncture technique and added to the study as engaged research investigators. The Food and Drug Administration (FDA) regulates acupuncture needles as a class II medical device, because they are intended for use in the cure, mitigation, treatment, or prevention of disease in man or are intended to affect the structure or function of the body of man. The FDA regulates the acupuncture needles (see 21 CFR 880.5580). The needles being used are Hwato 0.30X100mm Acupuncture needles, which are exempt from premarket notification by the FDA for use in acupuncture and will be used in accordance with their FDA approved labeling.

ELIGIBILITY:
***THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.***

Inclusion Criteria:

* Male and female DoD beneficiaries, age 18 years or older,
* Diagnosed with medial tibial stress syndrome (in one or both of their lower extremities) OR subjects meeting criteria of pain in the posteromedial tibia with exercise and direct palpation of the posteromedial tibia. Subjects with acute and chronic diagnoses will be included.

Exclusion Criteria:

* Pregnant
* Any of the following in the lower extremity being included into the study:
* Active cellulitis of lower extremity
* Tibial stress fracture
* If they have ever had any prior acupuncture for medial tibial stress syndrome using the defined KB-2 points.
* Use of anticoagulants
* Neurologic deficits, to include abnormal sensation, hypo- or hyper-active reflexes, muscle weakness not attributable to pain
* History of needle-shock with acupuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Change in pain over time as measured by 11-point numerical pain rating score (NPRS-11) | Visit 1 (Day 1) Beginning, Visit 1 (Day 1) End, Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 12)
  The NPRS is a validated segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The common format is a horizontal bar or line.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). The NPRS can be administered verbally (therefore also by telephone) or graphically for self-completion.
Change in pain over time as measured by Pain Disability Index (PDI) | Visit 1 (Day 1) , Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 12)
  The PDI score is a measure of functional status incorporating the dimensions of family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life support activities. The total of these dimensions provides the PDI score, which has been studied as clinically significant when a decrease of 9 points was observed. A score of 0 means no disability at all, and a score of 10 signifies that all of the activities in which you would normally be involved have been totally disrupted or prevented by the patient's pain.

SECONDARY OUTCOMES:
Change in Medial Tibial Stress Syndrome (MTSS) Score over time | Visit 1 (Day 1) , Visit 2 (Week 2), Visit 3 (Week 4), Visit 4 (Week 12)
  This a score of patient-related outcome measures. Score ranges from 0 (no limitation) to 10 (full limitation). The MTSS score specifically measures pain experienced along the shin and limitations due to shin pain. For the purpose of this study, we will compare the MTSS score reduction to NPRS-11 and look for a concurrent MTSS score decrease by 2 for clinical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Creech, DO, Principal Investigator — Eglin AFB, United States Air Force
Locations (1):
- 96th Medical Group, Eglin Air Force Base, Florida, United States

REFERENCES:
- [Background] Garnock C, Witchalls J, Newman P. Predicting individual risk for medial tibial stress syndrome in navy recruits. J Sci Med Sport. 2018 Jun;21(6):586-590. doi: 10.1016/j.jsams.2017.10.020. Epub 2017 Oct 23. PMID 29122474
- [Background] Winters M, Eskes M, Weir A, Moen MH, Backx FJ, Bakker EW. Treatment of medial tibial stress syndrome: a systematic review. Sports Med. 2013 Dec;43(12):1315-33. doi: 10.1007/s40279-013-0087-0. PMID 23979968
- [Background] Rompe JD, Cacchio A, Furia JP, Maffulli N. Low-energy extracorporeal shock wave therapy as a treatment for medial tibial stress syndrome. Am J Sports Med. 2010 Jan;38(1):125-32. doi: 10.1177/0363546509343804. Epub 2009 Sep 23. PMID 19776340
- [Background] Reshef N, Guelich DR. Medial tibial stress syndrome. Clin Sports Med. 2012 Apr;31(2):273-90. doi: 10.1016/j.csm.2011.09.008. PMID 22341017
- [Background] Soer R, Reneman MF, Vroomen PC, Stegeman P, Coppes MH. Responsiveness and minimal clinically important change of the Pain Disability Index in patients with chronic back pain. Spine (Phila Pa 1976). 2012 Apr 15;37(8):711-5. doi: 10.1097/BRS.0b013e31822c8a7a. PMID 21796022